CLINICAL TRIAL: NCT01167036
Title: Immediate Effectiveness of Instrument Assisted Soft Tissue Mobilization Compared to Placebo on the Sensitivity of Latent Upper Trapezius Trigger Points: A Randomized Double Blind, Placebo-controlled, Parallel-group Study
Brief Title: Effectiveness of a Massage Instrument Compared to Placebo for Upper Trapezius Muscle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglo-European College of Chiropractic (Other)
Responsible Party: Hugh Gemmell Principal Lecturer, Anglo-European College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AECC 20091
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-08

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial pain syndrome; Trigger points, Myofascial; Chiropractic; Massage; Musculoskeletal manipulation
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FascialEdge tool (Experimental): A massage tool used to loosen adhesions in the superficial fascia
  Interventions: Device: FascialEdge instrument
- Placebo (Placebo Comparator): Detuned electric point stimulation over the upper trapezius trigger point
  Interventions: Other: Placebo electric point stimulation

INTERVENTIONS:
Device: FascialEdge instrument — Stroking massage to patient tolerance over the muscle
  Other Names: FascialEdge tool
  Arms: FascialEdge tool
Other: Placebo electric point stimulation — Detuned electric point stimulation over the involved muscle
  Other Names: Pointer Plus stimulator
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine if using a specialized massage tool was more effective than a placebo treatment in relieving pain in the upper trapezius muscle along the top of the shoulder.

DETAILED DESCRIPTION:
The purpose of the study was to determine if a statistically significant and clinically meaningful difference exits between the FascialEdge tool and placebo in the treatment of latent upper trapezius trigger points.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* between 18-64 years of age
* a latent trigger point of the upper trapezius muscle

Exclusion Criteria:

* an active trigger point of the upper trapezius muscle
* rash or infection of the skin over the trigger point
* neck pain
* taking anticoagulant drugs
* spontaneous bleeding
* long term corticosteroid use

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold over the upper trapezius muscles as determined with a pressure pain algometer | Within five minutes after initial and only treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Gemmell, DC, EdD, Principal Investigator — Anglo-European College of Chiropractic
Locations (1):
- Anglo-European College of Chiropractic, Bournemouth, Dorset, United Kingdom